CLINICAL TRIAL: NCT00963781
Title: A Clinical Evaluation of Dual Antiplatelet Therapy Duration Following Treatment With the Medtronic Endeavor Zotarolimus-eluting Coronary Stent
Brief Title: Scripps Evaluation of Antiplatelet Therapies for Intermediate Duration With the Endeavor Stent (Seaside)
Acronym: SEASIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scripps Health (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Paul S Teirstein, MD, Director, Scripps Cardiovascular Institute, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-5248
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease; Coronary Thrombosis
Keywords: Coronary Artery Disease; Drug-Eluting Stents; Coronary Thrombosis; Platelet Aggregation Inhibitors; Coronary Restenosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Thrombosis; Coronary Restenosis | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Six months DAPT (Experimental): All patients will be assigned to 6 months of DAPT
  Interventions: Device: Medtronic Endeavor Stent; Drug: Reduced duration (6 months) DAPT

INTERVENTIONS:
Device: Medtronic Endeavor Stent — The study population was to consist of 900 consecutive, eligible patients with ischemic heart disease scheduled to undergo elective percutaneous coronary revascularization and amenable to treatment with an Endeavor drug-eluting stent with reference vessel diameter between 2.5 and 4.0 mm. Patients will be assigned to 6 month duration of post-procedure thienopyridine treatment with indefinite aspirin (minimum 81 mg daily) according to protocol. Recruitment was terminated early due to difficulty recruiting patients and difficulty achieving patient compliance with the six month anti-platelet protocol.
Drug: Reduced duration (6 months) DAPT

SUMMARY:
Despite the benefit of drug-eluting stents (DES) to reduce the need for repeat revascularization procedures, concerns regarding late stent thrombosis (ST) have led to recent guidelines advocating extended prescription of dual antiplatelet therapy (DAPT) with aspirin and a thienopyridine (clopidogrel or ticlopidine]) beyond that described in the product labeling. Specifically, an advisory has recommended at least 1 year DAPT following treatment with DES in patients without contraindications. However, this recommendation was largely empiric and not based on any trial showing reductions in ST with long-term DAPT, nor are potential safety differences between DES considered. Further, no study has examined the balance in potential efficacy with long-term DAPT relative to an increased bleeding risk.

A consistency across clinical trials involving the Endeavor DES has been very low rates of late myocardial infarction, cardiac death and ST. Unlike other DES, recent studies indicate that the Endeavor stent may permit more rapid and complete healing over stent struts in addition to restoring normal blood vessel function. Further, in patients treated with the Endeavor stent, long-term safety outcomes are similar through 3 years follow-up irrespective of whether patients were adherent to DAPT for durations of ≤ 6 months, 12 months or 24 months.

In this study, long-term safety and effectiveness will be examined for patients treated with the Endeavor stent and assigned to DAPT for reduced duration of 6 months. If the study demonstrates safety and efficacy, it could influence treatment guidelines in favor of an abbreviated duration of DAPT for patients treated with the Endeavor stent. This would mean that should a bleeding complication or need or surgery arise less than 12 months post-PCI, patients treated with the Endeavor stent could stop DAPT after 6 months with reasonable estimate of safety. Furthermore, it is possible that patients who are currently denied DES due to known need for elective surgery could be treated with the Endeavor stent in cases where surgery can be temporarily delayed. Finally, it could be an additional option for patients who forgo treatment with DES in favor of bare metal stent (BMS) out of fear of possible bleeding with long-term DAPT.

Finally, it is recognized that not all patients respond the same way to anti-platelet therapy. Recent studies have indicated that inherited genetic variations in the way the body metabolizes anti-platelet medications may be important determinants of responsiveness to thienopyridine therapy, and that such differences may also confer a higher likelihood of adverse outcome. Patients agreeing to the additional genetic sub-study will have a DNA sample taken at baseline to test for the presence of such genes related to antiplatelet therapy metabolism and effectiveness. The results of these tests could help the medical community to better understand individual variation in response to anti-platelet therapy and the role that genetics may play in determining the response. It is possible that the information gained could help physicians tailor DAPT on a patient by patient basis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is > 18 years of age.
2. The patient must be reliable, cooperative and willing to comply with all protocol-specified procedures and follow-up
3. The patient has clinical evidence of ischemic heart disease, stable or unstable angina, silent ischemia, or a positive functional study.
4. The patient has at least one lesion ≥50% diameter stenosis (de novo and/or restenotic, including in-stent bare metal stent restenosis) within a native coronary artery or bypass graft requiring percutaneous revascularization with stenting. (Note: Measurements may be made by careful visual estimate, on-line quantitative coronary angiography or intravascular ultrasound [IVUS].)
5. The target lesion(s) reference vessel diameter is 2.5 to 4.0 mm
6. The patient is an acceptable candidate for PTCA, stenting, and emergent coronary artery bypass grafting (CABG) surgery.
7. Female patients of childbearing potential must have a negative pregnancy test within 7 days before the procedure.
8. The patient or patient's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the enrolling clinical site.

Exclusion Criteria:

1. Planned treatment for any of the following patient and/or lesion characteristics:

   * Unprotected left main disease
   * Stage 4 chronic kidney disease, defined as creatinine clearance <30 mL/min and/or hemodialysis
   * Planned 2-stent treatment of a bifurcation lesion
   * Lesion length >30 mm
   * Lesion containing angiographic evidence of thrombus
   * Treatment of 3 vessel coronary disease
   * Severe left ventricular dysfunction (<25%)
   * In-stent restenosis of previously placed DES
2. A known hypersensitivity or contraindication to cobalt, nickel, chromium, molybdenum, polymer coatings (e.g., phosphorylcholine), or a sensitivity to contrast media, which cannot be adequately pre-medicated.
3. History of an allergic reaction or significant sensitivity to drugs such as zotarolimus, rapamycin, tacrolimus, everolimus, or any other analogue or derivative.
4. A known hypersensitivity to clopidogrel, ticlopidine, aspirin, heparin or bivalirudin. Note: allergy to one thienopyridine type, but not another, does not constitute an exclusion.
5. A platelet count < 100,000 cells/mm³ or > 700,000 cells/mm³, or a white blood cell (WBC) count < 3,000 cells/mm³.
6. Evidence of recent/acute MI/acute coronary syndrome within preceding 6 months of the intended index procedure (defined as: dynamic ST-segment/T wave electrocardiographic changes and/or Q wave myocardial infarction (QWMI) or non-Q wave myocardial infarction (NQWMI) having CK enzymes > 2X the upper laboratory normal with the presence of a CK-MB elevated above the Institution's upper limit of normal, or troponin level elevated above the Institution's upper limit of normal).
7. Treatment within the target vessel with any stent type within the previous 9 months
8. Prior to procedure, intended use of DES other than Endeavor stent
9. Active peptic ulcer or upper gastrointestinal (GI) bleeding within the prior 6 months.
10. History of bleeding diathesis or coagulopathy or patient will refuse blood transfusions.
11. Concurrent medical condition with a life expectancy of less than 12 months.
12. Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study.
13. Currently participating in an investigational drug or another device study that clinically interferes with the current study endpoints
14. Inability to comply with protocol required medication regimen (eg, [minimum] 6 month protocol-specified dual antiplatelet duration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2009-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of all-cause death/myocardial infarction (MI)/stroke/definite and probable stent thrombosis (ST) at 1 year post-procedure (Hierarchal) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David E Kandzari, MD, Principal Investigator — Scripps Clinic; Paul S. Teirstein, MD, Principal Investigator — Scripps Clinic; Eric J. Topol, MD, Principal Investigator — Scripps Clinic and Scripps Translational Science Institute
Locations (1):
- Scripps Clinic, La Jolla, California, United States